CLINICAL TRIAL: NCT00521014
Title: A Phase II Study of GM-CSF (Sargramostim) and Rituximab Following Autologous Transplantation For Relapsed Follicular Lymphoma
Brief Title: GM-CSF and Rituximab After Autologous Stem Cell Transplant in Treating Patients With Relapsed or Refractory Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-085; P30CA008748 (NIH); MSKCC-07085; BRLX-MSKCC-07-085
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Filgrastim; Rituximab; sargramostim; Carmustine; Cytarabine; Etoposide; Melphalan

ARMS (1):
- GM-CSF and Rituximab After Autologous Stem Cell Transplant (Experimental): GM-CSF: 250 mcg (flat dose) three times per week for 8 weeks, administered on alternate days. Thus, 24 doses of GM-CSF will be administered.
  Rituximab: 375 mg/m2/week for 4 weeks, beginning within 3 days after the first dose of GM-CSF; rituximab. The second course of GM-CSF and rituximab will be administered approximately 22-26 weeks (day +154 to +182) after ASCT.
  Interventions: Biological: filgrastim; Biological: rituximab; Biological: sargramostim; Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Biological: sargramostim
Drug: carmustine
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Procedure: autologous hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving high-dose chemotherapy before an autologous stem cell transplant helps stop the growth of cancer cells by stopping them from dividing or by killing them. An autologous stem cell transplant may be able to replace the blood-forming cells that were destroyed by chemotherapy. GM-CSF may increase the number of immune cells found in bone marrow or peripheral blood. Giving a monoclonal antibody, such as rituximab, after the transplant may find any remaining cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Giving GM-CSF together with rituximab after autologous stem cell transplant may be an effective treatment for follicular non-Hodgkin lymphoma.

PURPOSE: This phase II trial is studying how well giving GM-CSF together with rituximab after autologous stem cell transplant works in treating patients with relapsed or primary refractory follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the progression-free survival rate at 2 years after autologous stem cell transplantation (ASCT) in patients with relapsed or primary refractory follicular lymphoma treated with sargramostim (GM-CSF) and rituximab after ASCT.

Secondary

* To assess the safety of administering GM-CSF and rituximab after ASCT.
* To assess the effects of GM-CSF on the relative expression of activating and inhibitory FcγR on circulating monocytes.
* To assess the effects of GM-CSF on the relative expression of activating and inhibitory FcγR on circulating dendritic cells.
* To assess the effects of GM-CSF on the level of circulating FcγR.
* To assess the reconstitution of NK cells, NK-T cells, dendritic cell subsets, and regulatory T-cells after ASCT.

OUTLINE:

* High-dose chemotherapy: Patients receive carmustine IV over 2 hours on day -7, etoposide IV over 1 hour and cytarabine IV every 12 hours on days -6 to -3, and melphalan IV on day -2.
* Autologous stem cell transplantation (ASCT): Patients undergo ASCT on day 0. Patients receive filgrastim (G-CSF) subcutaneously (SC) once a day beginning on day 5 and continuing until blood counts recover.
* Sargramostim (GM-CSF) and rituximab: Beginning approximately 7-10 weeks (49-70 days) after ASCT, patients receive GM-CSF SC 3 times a week for 8 weeks and rituximab IV once weekly for 4 weeks (beginning within 3 days after the first dose of GM-CSF). Patients receive a second course of GM-CSF and rituximab (as above) beginning approximately 22-26 weeks (154-182 days) after ASCT.

After the completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic diagnosis of grade 1, 2, 3, or transformed follicular lymphoma
* Achieved a complete or partial response to last salvage therapy

  * Completed salvage therapy within the past 12 weeks
  * No disease progression since last salvage therapy
* One of the following disease statuses must have been present prior to receiving salvage therapy

  * Refractory to last anti-lymphoma therapy
  * Last remission duration less than 1½ years if salvage therapy is 3rd regimen
  * Last remission duration less than 3 years if salvage therapy is 2nd regimen
* Minimum of 2 x 10^6 CD34+ cells/kg cryopreserved and available for hematopoietic stem cell support
* No leptomeningeal disease or brain parenchyma involvement

PATIENT CHARACTERISTICS:

* Cardiac ejection fraction > 50%

  * If over 60 years of age, no evidence of cardiac ischemia by treadmill stress test (stress echo or sesta-MIBI)
* Adjusted diffusing capacity ≥ 50% of the predicted value on pulmonary function testing
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 50 mL/min
* ANC > 1,000/μL
* Platelet count > 50,000/μL
* Total bilirubin ≤ 2.0 mg/dL (≤ 3.0 mg/dL if Gilbert's disease is suspected)
* Not pregnant or breast-feeding
* Fertile patients must use an acceptable form of birth control
* HIV I or II negative
* No acute or chronic hepatitis B
* No active hepatitis C
* No medical illness (unrelated to non-Hodgkin lymphoma), including malignancies that, in the opinion of the attending physician and/or principal investigator, would preclude study treatment
* No other malignancy within the past 5 years except curatively treated cutaneous basal cell or squamous cell carcinoma or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* No more than 3 prior anti-lymphoma regimens, inclusive of the salvage therapy

  * Biologic agents (e.g., monoclonal antibodies and vaccines) administered as part of a planned treatment regimen will not be considered distinct regimens
  * Chemotherapy administered primarily for the purpose of stem cell mobilization (e.g., cyclophosphamide at 2-4 g/m²) will not be considered an anti-lymphoma regimen
* No prior autologous or allogeneic hematopoietic stem cell transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Matthew Matasar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Relapsed Follicular Lymphoma Patients: Study of GM-CSF (Sargramostim) and Rituximab Following Autologous Transplantation For Relapsed Follicular Lymphoma GM-CSF: 250 mcg (flat dose) three times per week for 8 weeks, Rituximab: 375 mg/m2/week for 4 weeks, beginning within 3 days after the first dose of GM-CSF
Period: Overall Study
Arm/Group | Relapsed Follicular Lymphoma Patients
Started | 14
Completed | 13
Not Completed | 1
Not completed — Inevaluable, not treated | 1

BASELINE CHARACTERISTICS:
Groups:
- Relapsed Follicular Lymphoma Patients: Study of GM-CSF (Sargramostim) and Rituximab Following Autologous Transplantation For Relapsed Follicular Lymphoma
Arm/Group | Relapsed Follicular Lymphoma Patients
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: after autologous stem cell transplantation (ASCT). Disease progression is defined using International Workshop Criteria for non-Hodgkin lymphoma37 and is defined as:
  1. ≥ 50% increase in products of diameters of any previously identified abnormal node or nodule AND/OR
  2. appearance of any new lesions
Time Frame: up to 3 years
Measure: Mean (Full Range); unit: years
Arm/Group | Relapsed Follicular Lymphoma Patients
Number analyzed (Participants) | 13
years | 1.759 [0.47 to 2.3]

ADVERSE EVENTS:
Arm/Group | Relapsed Follicular Lymphoma Patients
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Follicular Lymphoma Patients (N=13)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Inf norm ANC/gr1/2 (Infections and infestations) | 1 (1)
Obstruction, GI- Gallbladder (Gastrointestinal disorders) | 1 (1)
Pain - Buttock (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed Follicular Lymphoma Patients (N=13)
ALT, SGPT (Blood and lymphatic system disorders) | 5 (5)
AST, SGOT (Blood and lymphatic system disorders) | 2 (2)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1)
Amylase (Blood and lymphatic system disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (6)
Hemoglobin (Blood and lymphatic system disorders) | 13 (13)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13 (13)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 13 (13)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 10 (10)
Platelets (Blood and lymphatic system disorders) | 13 (13)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes